CLINICAL TRIAL: NCT06515483
Title: Evaluation of the Efficacy and Safety of a Loop Stretchable Dental Floss in Controlling Gingivitis and Supragingival Plaque Removal During Thirty Days
Brief Title: Evaluation of the Efficacy and Safety of a Loop Stretchable Dental Floss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ana G. Gossweiler, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22752
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-02

CONDITIONS: Gingivitis; Supragingival Plaque
Keywords: Dental floss, gingivitis, plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: A sufficient number of subjects will be screened to participate, and 64 will be randomized. We intend to randomize a nearly equal number of female and male subjects. A unique screening number will identify all subjects screened for study participation. Screening numbers will be assigned according to appearance at the study site. Subjects who meet all inclusion and exclusion criteria will be randomized into the study. Block randomization will be used to assign subjects to one of the two sequences: control regiment or experimental regimen. Randomization will be stratified by gender. Randomization numbers will be assigned using randomization schedules provided by the IU Department of Biostatistics and Health Data Science statistician.
Who Masked: Outcomes Assessor
Masking Description: The clinical examiner will remain blind to the individual subjects' treatment group during the entire study. If the treatment assignment must be unblinded for a subject, such as in the case of an emergency, the Investigator will provide written documentation of the unblinding request. Unblinding would involve withdrawing the subject from the study. Otherwise, blinding will not be broken, unless required in the circumstances detailed above, until all subjects have completed the final study visit and the database has been monitored, locked, and approved by the Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 (Experimental): Brushing and Flossing
  Interventions: Device: Brushing and Flossing of teeth
- Arm 2 (Placebo Comparator): Brushing only
  Interventions: Other: Brushing Only

INTERVENTIONS:
Device: Brushing and Flossing of teeth — 32 subjects will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects in the experimental group will brush and floss with the provided stretchable loop floss at least twice a day. To assess compliance, each subject will be asked to fill out a diary every time they brush/floss. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.
  Arms: Arm 1
Other: Brushing Only — 32 subjects will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects assigned to the control group will brush their teeth at least twice a day only. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.
  Arms: Arm 2

SUMMARY:
This will be a single-blind, single-center, parallel, randomized controlled clinical trial to evaluate the efficacy and safety of Floss Loops stretchable floss for the control of gingivitis and supragingival plaque removal between two groups, control (no-floss) and experimental (flossing with Floss Loops), during thirty (2 +/-) days.

DETAILED DESCRIPTION:
At the screening/baseline visit, potential subjects will be given the IRB-approved informed consent form to read and ask questions. After the subject signs and dates the consent, the study representative will sign and date the consent to confirm that the consent process was completed before initiating any study procedures. The subject will be given a copy of the signed consent. The study dentist will collect and review information related to the subject's demographic, medical, and concomitant medications. The subject will have a hard and soft tissue exam, as well as a clinical examination of the gums and dental plaque present using the Lobene modified gingival index for gingivitis assessment, the marginal bleeding on probing index and the Turesky modification of the Quigley and Hain plaque index.

A total of 64 subjects who meet the study criteria will be enrolled and randomized into two groups. 32 subjects will be assigned to the control group (Brushing twice a day only and no flossing) and 32 to the experimental group (Brushing and Flossing with the stretchable loop floss twice daily). Each subject will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects assigned to the control group will brush their teeth at least twice a day only, and subjects in the experimental group will brush and floss with the provided stretchable loop floss at least twice a day. To assess compliance, each subject will be asked to fill out a diary every time they brush/floss. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.

All clinical examinations will be performed by examiners who will be blind to the subject's oral hygiene procedures.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male subjects between 18 to 65 years old
* Willing to read and sign the IRB-approved informed consent
* Healthy, as determined by pertinent medical history at the examiner dentist's discretion
* A minimum of 20 natural teeth (excluding third molars) with at least two scorable surfaces per tooth (teeth with full crowns, large/extensive restorations on the interproximal areas, and orthodontic bands will not be included in the tooth count)
* Mild to moderate plaque and gingivitis GI of 1.75 or greater (The Lobene-modified gingival index score) calculation made based on a whole mouth score
* PLI of 1.95 or greater (Turesky modification of the Quigley and Hein Plaque Index) calculation based on a whole mouth plaque score
* Be willing to comply with study visits and requirements

Exclusion Criteria:

* Presence of any acute or chronic condition, organ system disease, or medication that, in the principal investigator's opinion, could compromise the subjects' ability to participate in the study
* Gross oral pathologies, including caries, calculus, or soft tissue conditions that show evidence of chronic neglect
* Orthodontic appliances appliances (except for fixed lingual retainers, teeth will be excluded from the teeth count) or any removable prosthesis
* Evidence of acute periodontal conditions or periodontitis with pockets greater than 5 mm on more than one site
* Taking antibiotics two weeks before baseline procedures and throughout the study
* Need for antibiotic prophylaxis prior to dental procedures
* Use of daily anti-inflammatory drugs (NSAID, TNF- AB, others) within 30 days before baseline
* Pregnant, wanting to get pregnant, or breast-feeding female
* Acute Temporomandibular Disorders (TMD)
* Subject who has participated in other studies (including non-medicinal studies) involving product(s) within 30 days before study entry
* Subject who has previously been randomized in this study
* Self-reported allergy to disclosing solution ingredients (red dye #28)
* An employee of the study site directly involved with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana G Gossweiler, DDS/MSD, Principal Investigator — Indiana University School of dentistry, Oral Health Research Institute
Locations (1):
- Indiana University School of dentistry, Oral Health Research institute 415 Lansing Street, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotsakis GA, Lian Q, Ioannou AL, Michalowicz BS, John MT, Chu H. A network meta-analysis of interproximal oral hygiene methods in the reduction of clinical indices of inflammation. J Periodontol. 2018 May;89(5):558-570. doi: 10.1002/JPER.17-0368. PMID 29520910
- [Background] Shamsoddin E. Dental floss as an adjuvant of the toothbrush helps gingival health. Evid Based Dent. 2022 Sep;23(3):94-96. doi: 10.1038/s41432-022-0818-x. Epub 2022 Sep 23. PMID 36151277
- [Background] Alali AY, Al-Khabbaz A, Michael S, Swain MV. Frictional coefficient during flossing of teeth. Dent Mater. 2018 Dec;34(12):1727-1734. doi: 10.1016/j.dental.2018.09.002. Epub 2018 Sep 21. PMID 30244840
- [Background] Huang Z, Broadbent JM, Choi JJE. Comparison of dental flosses - an investigation of subjective preference and mechanical properties. Biomater Investig Dent. 2023 Sep 22;10(1):2258919. doi: 10.1080/26415275.2023.2258919. eCollection 2023. PMID 37753304
- [Background] Carr MP, Rice GL, Horton JE. Evaluation of floss types for interproximal plaque removal. Am J Dent. 2000 Aug;13(4):212-4. PMID 11763934
- [Background] Rich SK, Friedman JA, Schultz LA. Effects of flossing on plaque and gingivitis in third grade schoolchildren. J Public Health Dent. 1989 Spring;49(2):73-7. doi: 10.1111/j.1752-7325.1989.tb02029.x. PMID 2709366
- [Background] Azcarate-Velazquez F, Garrido-Serrano R, Castillo-Dali G, Serrera-Figallo MA, Ganan-Calvo A, Torres-Lagares D. Effectiveness of flossing loops in the control of the gingival health. J Clin Exp Dent. 2017 Jun 1;9(6):e756-e761. doi: 10.4317/jced.53858. eCollection 2017 Jun. PMID 28638551
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Londero AB, Reiniger APP, Tavares RCR, Ferreira CM, Wikesjo UME, Kantorski KZ, Moreira CHC. Efficacy of dental floss in the management of gingival health: a randomized controlled clinical trial. Clin Oral Investig. 2022 Aug;26(8):5273-5280. doi: 10.1007/s00784-022-04495-w. Epub 2022 Apr 22. PMID 35451656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on October 15 and ended on December 4th. Recruitment was conducted in the OHRI Clinic.
Pre-assignment Details: There were not significant events reported prior to participants enrollment.
Groups:
- Brushing and Flossing: 32 subjects were instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects in the experimental group brushed and flossed with the provided stretchable loop floss at least twice a day. To assess compliance, each subject was asked to complete a diary every time they brushed or flossed. On day 15 (+/- 2) day of product use, subjects received a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction applied, and the efficacy assessments were repeated, subjects were dismissed, and the study was finished.
- Brushing Only: 32 subjects were instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects assigned to the control group brushed their teeth at least twice a day only. On day 15 (+/- 2) day of product use, subjects received a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction applied, and the efficacy assessments were repeated, subjects were dismissed, and the study was finished.
Period: Overall Study
Arm/Group | Brushing and Flossing | Brushing Only
Started (1. Subject's received a phone call 15 days after baseline visit for compliance assessment and remind subjects of 30 days appointment 2. Subjects end of treatment period visit that occurred 30 days after baseline visit.) | 32 (All participants in this group received a phone call at the 15 day (+-2 day) for compliance assessment. 1 subject withdrew at the time of the 15-day call due to family issues and did not participate in the final visit.) | 32 (All participants in this group received a 15 day (+-2 day) compliance assessment phone call and all of them participated on the final visit assessments.)
Completed | 31 (1 subject was lost to follow up) | 32
Not Completed | 1 | 0
Not completed — Subject withdraw due to family issues | 1 | 0

BASELINE CHARACTERISTICS:
Population: Both groups had 32 participants at the beginning of the study.
Groups:
- Brushing and Flossing: Brushing and Flossing
  Brushing and Flossing of teeth: 32 subjects will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects in the experimental group will brush and floss with the provided stretchable loop floss at least twice a day. To assess compliance, each subject will be asked to fill out a diary every time they brush/floss. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.
- Brushing Only: Brushing only
  Brushing Only: 32 subjects will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects assigned to the control group will brush their teeth at least twice a day only. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.
- Total: Total of all reporting groups
Arm/Group | Brushing and Flossing | Brushing Only | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 43.225 [19 to 63] | 42.36 [21 to 63] | 42.792 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64
The Modified Gingival Index by Lobene [Mean (Standard Deviation); unit: Index] — The Lobene-modified gingival index was access by evaluating each tooth on six surfaces (Mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). Each surface was scored based on the inflammatory visual changes, severity, and extent. A score would range from 0.1 to 3.0 (0.1-1.0= = mild inflammation; 1.1-2.0= = moderate inflammation; and 2.1-3.0= = severe inflammation). For the MGI calculation over all and interproximal, all the values for each tooth were added and divided by the number of surfaces examined.
  Index | 2.335 (0.047) | 2.257 (0.042) | 2.296 (0.032)
Bleeding on Probing [Mean (Standard Deviation); unit: Percentage of bleeding sites] — BOP was assessed at the Mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual surfaces. A periodontal probe was inserted into the gingival crevice at an angle of approximately 60°. BOMP was read up to 30 seconds after probing. The surfaces were scored as negative (0=no ) or positive (1). The percentage of bleeding sites was determined by adding up the number of bleeding sites, divided by the total number of probing sites, and multiplying by 100. Percentage of Bleeding sites between 20% 40 are considered moderate. Below 20% mild and higher than 40%severe.
  Percentage of bleeding sites | 25.18 (2.27) | 24.87 (2.35) | 25.03 (1.62)
Turesky Dental Plaque Index [Mean (Standard Deviation); unit: Index] — Each tooth, except the third molars, was scored on six sites (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). The scores would range from 0 (No plaque) to 5 (Plaque covering 2/3 of the crown or more). The plaque score index for an individual was determined by adding all the individual scores and dividing the total score by the number of surfaces examined. Scores o to 2 are considered mild, scores 2 to 3 moderate and higher that 3 high.
  Index | 4.026 (0.063) | 3.947 (0.061) | 3.986 (0.044)

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Assessment
Description: Dental plaque was identified using a disclosing solution and scored using the Turesky modification of the Quigley-Hein Plaque Index (PLI). The index score was scored between 0 and 5, with 0 = no plaque detected and 5= = Plaque covering 2/3 or more of the tooth's crown. The remaining values are based on the amount of plaque covering the tooth. The higher the score, the more plaque accumulated and the worse the outcome for the surface. Each tooth, except the third molars, will be scored at six sites: Mesio-Buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual. The plaque score index for an individual is determined by adding all the individual scores and dividing the total score by the number of surfaces examined.
Time Frame: Baseline and 30 days examination
Population: One patient who did not complete the 30-day follow-up examination was not included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Brushing and Flossing: Brushing and Flossing of teeth: 32 subjects will be instructed to clean their teeth daily using only the provided toothbrush with an assigned ADA-accepted fluoride dentifrice. Subjects in the experimental group will brush and floss with the provided stretchable loop floss at least twice a day. To assess compliance, each subject will be asked to fill out a diary every time they brush/floss. On day 15 (+/- 2) day of product use, subjects will receive a phone call from the study coordinator or designee to assess brushing/flossing compliance. At day 30 (+/- 2), study hygiene and gum chewing restrictions as well as eating restriction will apply, and the efficacy assessments will be repeated, subjects will be dismissed, and the study will finish.
Arm/Group | Brushing and Flossing | Brushing Only
Number analyzed (Participants) | 31 | 32
Index
  Baseline | 4.026 (0.063) | 3.947 (0.061)
  30 days | 3.856 (0.036) | 3.892 (0.047)
  PLI change from baseline to 30 days | -0.170 (0.046) | -0.055 (0.057)
Statistical Analysis 1: Comparison: Brushing and Flossing vs Brushing Only; Due to non-normally distributed data, differences in each index between the experimental and control groups at baseline were compared using non-parametric Wilcoxon Rank Sum tests; Test type: Other; p = 0.323, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.095 to 0.254] — Comparing baseline PLI between groups
Statistical Analysis 2: Comparison: Brushing and Flossing vs Brushing Only; Due to non-normally distributed data, differences in each index between the experimental and control groups at 30 days were compared using non-parametric Wilcoxon Rank Sum tests; Test type: Other; p = 0.371, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -0.036, 95% CI 2-sided [-0.156 to 0.084] — Comparing 30-day PLI between groups
Statistical Analysis 3: Comparison: Brushing and Flossing vs Brushing Only; Test type: Other; p = 0.120, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Net) = -0.115, 95% CI 2-sided [-0.262 to 0.031] — Comparing the mean difference in PLI from baseline to 30 days between groups

2. Primary Outcome: Gingivitis Assessment
Description: The Lobene-modified gingival index (MGI) will be used. This is a non-invasive index that assesses the health of the gums based on their visual clinical appearance. Each tooth will be evaluated visually on six surfaces (Mesio-buccal, buccal, distobuccal, mesio-lingual, lingual, and disto-lingual). Each surface will be scored based on the inflammatory visual changes, severity, and extent. For the MGI calculation, all the values for each tooth will be added and divided by the number of surfaces examined. Scores range from 0 to 4. A score of 0 will represent normal. A score of 1 and 2 will represent mild inflammation, a score of 3 indicates moderate inflammation and a score of 4 indicates severe inflammation). A single, trained examiner will complete all the examinations.
Time Frame: Baseline and 30 days examination
Population: One patient who did not complete the 30-day follow-up examination was not included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Brushing and Flossing | Brushing Only
Number analyzed (Participants) | 31 | 32
Index
  Baseline | 2.335 (0.047) | 2.257 (0.042)
  30 days | 2.227 (0.049) | 2.312 (0.033)
  MGI change from baseline to 30 days | -0.108 (0.031) | 0.055 (0.030)
Statistical Analysis 1: Comparison: Brushing and Flossing vs Brushing Only; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.270, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [-0.048 to 0.204] — Comparing baseline MGI between groups
Statistical Analysis 2: Comparison: Brushing and Flossing vs Brushing Only; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.071, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -0.085, 95% CI 2-sided [-0.203 to 0.033] — Comparing 30-day MGI between groups
Statistical Analysis 3: Comparison: Brushing and Flossing vs Brushing Only; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -0.163, 95% CI 2-sided [-0.249 to -0.077] — Comparing the mean difference in MGI from baseline to 30 days between groups

3. Secondary Outcome: Bleeding on Marginal Probing (BOMP)
Description: Bleeding on probing will be assessed at six surfaces (Mesio-buccal, buccal, distobuccal, mesio-lingual, lingual, and disto-lingual). A periodontal probe with a rounded tip 0.5mm in diameter will be gently inserted into the gingival crevice to a depth of approximately 2 mm and run at an angle of roughly 60° about the longitudinal axis of the tooth, except for third molars if present. BOPBOMP will be read up to 30 seconds after probing. The surfaces would be scored as negative (0=no BOPBOMP) or positive (1=BOPBOMP). The whole-mouth BOPBOMP score will be calculated as the percentage of bleeding sites, will be determined by adding up the number of bleeding sites, dividing this number by the total number of probing sites, and multiplying by 100. Percentage of Bleeding sites between 20% 40 are considered moderate. Below 20% mild and higher than 40%severe.
Time Frame: Baseline and 30 days examination
Population: One patient who did not complete the 30-day follow-up examination was not included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Percentage of bleeding sites
Arm/Group | Brushing and Flossing | Brushing Only
Number analyzed (Participants) | 31 | 32
Percentage of bleeding sites
  Baseline | 25.18 (2.27) | 24.87 (2.35)
  30 days | 17.41 (3.20) | 25.63 (2.62)
  BOMP change from baseline to 30 days | -7.77 (2.91) | 0.76 (2.59)
Statistical Analysis 1: Comparison: Brushing and Flossing vs Brushing Only; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.902, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-6.23 to 6.85] — Comparing baseline BOMP between groups
Statistical Analysis 2: Comparison: Brushing and Flossing vs Brushing Only; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -8.22, 95% CI 2-sided [-16.46 to 0.02] — Comparing 30-day BOMP between groups
Statistical Analysis 3: Comparison: Brushing and Flossing vs Brushing Only; Test type: Other; p = 0.032, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Net) = -8.53, 95% CI 2-sided [-16.31 to -0.75] — Comparing the mean difference in BOMP from baseline to 30 days between groups

ADVERSE EVENTS:
Time Frame: Adverse events for each subject were collected for 30 days. Starting at the baseline visit and ending at the time of the last visit (30 day visit)
Description: The definition did not differ. Adverse event information was collected by phone on day 15 and in person during the 30-day visit. No SAEs were reported during the study.
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

LIMITATIONS AND CAVEATS:
There were not limitations or caveats between the PI and the sponsor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT06515483/Prot_SAP_000.pdf